CLINICAL TRIAL: NCT06957418
Title: The Alzheimer's Disease Tau Platform Clinical Trial
Brief Title: Alzheimer's Tau Platform: Master Protocol
Acronym: ATP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paul S. Aisen (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, San Francisco (Other); Massachusetts General Hospital (Other); Alzheimer's Therapeutic Research Institute (Other); Alzheimer's Clinical Trials Consortium (Other)
Responsible Party: Sponsor-Investigator, Paul S. Aisen, Director, ATRI, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-014; R01AG078457 (NIH)
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Preclinical Alzheimer's Disease; Alzheimer Disease; Prodromal Alzheimer's Disease
Keywords: Alzheimer's disease; Preclinical Alzheimer's; Prodromal Alzheimer's; Mild cognitive impairment (MCI); Neurodegeneration; Dementia; Tau-directed therapy; Monoclonal antibody; Anti-tau therapy; Combination therapy; Immunotherapy; anti-amyloid mAb
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Nerve Degeneration; Dementia | interventions — AADvac1

STUDY DESIGN:
Intervention Model Description: As new investigational products become available, additional regimens will be added to the Alzheimer's Tau Platform trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A: AADvac1 (Experimental): Participants are randomized to receive either AADvac1, a tau directed monotherapy, combination AADvac1 with an anti-amyloid monoclonal antibody (mAb), or an anti-amyloid mAb alone (active control)
  Interventions: Drug: AADvac1
- Regimen B: Tau2 (Experimental): Participants are randomized to receive either Tau2 directed monotherapy, combination Tau2 directed therapy with an anti-amyloid monoclonal antibody (mAb), or an anti-amyloid mAb alone (active control)
  Interventions: Drug: Tau2

INTERVENTIONS:
Drug: AADvac1 — AADvac1 tau directed therapy
  Arms: Regimen A: AADvac1
Drug: Tau2 — Tau2 directed therapy
  Arms: Regimen B: Tau2

SUMMARY:
The goal of the Alzheimer's Tau Platform (ATP) is to evaluate the safety and effectiveness of tau-directed therapies, alone or in combination with an anti-amyloid monoclonal antibody (mAb), in adults aged 50-80 with late preclinical or early prodromal Alzheimer's disease.

This platform trial allows for the simultaneous testing of multiple tau therapies under a shared master protocol. This means that multiple investigational products will be tested simultaneously or sequentially. Each investigational product will be tested in a regimen.

The main questions the platform trial aims to answer are:

* Does any tau-directed therapy, alone or in combination with an anti-amyloid mAb, reduce brain tau deposition more than an anti-amyloid mAb, alone?
* Does any tau-directed therapy, alone or in combination with an anti-amyloid mAb, slow disease progression based on fluid biomarkers, imaging, or clinical measures?

Participants will:

* Be randomized to a treatment regimens, each containing different tau therapies. The exact number of treatment regimens that will active at the time of screening will change over time.
* Receive an anti-amyloid mAb or placebo for 6 months, followed by 24 months of tau therapy alone or in combination with an anti-amyloid mAb.
* Undergo regular cognitive testing, brain scans (MRI/PET), and biomarker assessments over 30 months

Participants will have an equal chance to be randomized to all regimens that are active at the time of screening. Once randomized to a regimen, participants will be randomized to one of three arms: (1) tau therapy alone, (2) a combination of an anti-amyloid mAb and tau therapy, or (3) an anti-amyloid mAb alone.

New regimens will be continuously added as new investigational products become available. The Alzheimer's Tau Platform Trial will enroll additional participants as each new regimen becomes available.

ATP is expected to launch with two regimens:

* Regimen A: AADvac1
* Regimen B: Tau2

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of the participant's informed consent to study procedures (including APOE genotyping).
2. Ages 50-80 years (inclusive). Participants between the ages of 50 and 60 (inclusive) must be mildly impaired at screening (global CDR=0.5 and maximum CDR-SB <1.5
3. Cognitively unimpaired (preclinical AD with a global CDR=0) or mildly impaired (prodromal AD with a global CDR=0.5 and maximum CDR-SB <1.5).
4. MMSE score at screening of 20-30 (inclusive) with educational adjustments:

   1. If <12 years of education, MMSE required to be >20.
   2. If 13 to 15 years (inclusive) of education, MMSE required to be >22.
   3. If >16 years of education, MMSE required to be >24.
5. Plasma biomarker result at screening that demonstrate the presence of amyloid pathology, consistent with preclinical-prodromal AD.
6. Elevated brain tau on PET (MTL or NEO tau SUVr >1.2) at screening.
7. Elevated brain amyloid on PET (centiloids > 40) at screening.
8. Stable doses of permitted medications as described per protocol for a minimum of 30 days prior to screening.
9. Resides at home or in the community (assisted living acceptable).
10. In the opinion of the site PI, has a study partner able and willing to provide accurate information (including clinical symptoms and medical history) about the participant and participate in study visits and informant-based assessments (usually requires at least 5 hours of contact per week) for the duration of the study.
11. As assessed by the site PI, participant is likely to be able to comply with the protocol for the duration of the study, and has adequate vision, hearing (hearing aid permitted), and literacy (English or Spanish) sufficient for compliance with the required testing procedures.
12. Must complete all screening evaluations as outlined per protocol.

Exclusion Criteria:

1. Females who are lactating or pregnant (as documented by a urine pregnancy test) during screening, or plan to become pregnant during the study.
2. Females of childbearing potential who did not use a highly effective method of contraception within 28 days of screening and/or are not willing to use highly effective method of contraception for the duration of their participation in the study. Males who are sexually active with a female of childbearing potential and do not agree to use barrier methods of contraception (condoms with spermicide) during the trial and for 6 months after the last dose of study drug unless the female is using a highly effective method of contraception.
3. Lacks good venous access such that multiple blood draws would be precluded.
4. Weighs less than 40kg, or more than 136kg at screening.
5. Suspected or known allergic reactions, adverse reactions, or hypersensitivity to any components of the study intervention for any of the available regimen.
6. Previous treatment with the study intervention from any available regimen unless it can be confirmed the participant received placebo in the previous study.
7. Prior or current treatment with a prohibited medication as described per protocol.
8. Enrollment in another investigational study as described per protocol. Participants enrolled in an observational study may be permitted with Medical Monitor review and approval.
9. Contraindications to MRI studies, including metal (ferromagnetic) implants, a cardiac pacemaker that is not compatible with MRI, and/or severe claustrophobia.
10. MRI scan at screening showing a single area of cerebral vasogenic edema, superficial siderosis, or showing more than four (4) cerebral microhemorrhages (defined as 10 mm or less at the greatest diameter); evidence of a prior or current macrohemorrhage (greater than 10 mm at greatest diameter, also referred to as intracerebral hemorrhage >1 cm within this protocol); cerebral contusion; encephalomalacia; aneurysms greater than 6 mm, or any aneurysms that have not been stable in size for the past 2 years; vascular malformations that are at high risk for hemorrhage; infectious lesions; evidence of multiple lacunar infarcts (that in the opinion of the investigator, may impact cognition); stroke involving a major vascular territory; severe small vessel disease; severe diffuse white matter disease; space occupying lesions; or brain tumors (however, lesions diagnosed as meningiomas or arachnoid cysts and less than 1 cm at their greatest diameter need not be exclusionary).
11. Contraindications to tau and/or amyloid PET scan imaging and/or use of MK6240 and/or 18F-NAV-4694 (flutafuranol).
12. For participants undergoing an LP as part of the optional longitudinal CSF biomarker sub-study, contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; international normalized ratio (INR) >1.4 or other coagulopathy; platelet count of <120,000/μL; infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of LP NOTE: low dose aspirin is permitted; degenerative arthritis of the lumbar spine; suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
13. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of study drug (e.g., moderate and/or severe untreated obstructive sleep apnea, clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular conditions), as per the site PI's judgement.
14. History of severe allergic reaction (e.g., anaphylaxis) including, but not limited to: severe allergic reaction to previous vaccines, foods, and/or medications.
15. Hospitalization within 30 days prior to screening or baseline.
16. Clinically significant infections or major surgical operation within 3 months prior to screening.
17. History of chronic or recurrent infections judged to be clinically significant by the site PI and which would potentially hamper the evaluation of efficacy and safety assessments.
18. Myocardial infarction within 1 year prior to baseline, unstable angina pectoris, or significant coronary artery disease.
19. History of cancer within the past 5 years other than treated squamous cell carcinoma, basal cell carcinoma and melanoma in-situ, in-situ prostate cancer, or in-situ breast cancer, which have been fully removed and are considered cured.
20. History of inflammatory neurological disorders.
21. History or presence of immunological or inflammatory conditions, including neurological disorders, judged to be clinically significant by the site PI.
22. History of meningitis or meningoencephalitis.
23. History of moderate or severe traumatic brain injury.
24. History or presence of uncontrolled seizures. If history of seizures, they must be well controlled with no occurrence of seizures in the 2 years prior to study screening. The use of antiepileptic medications is permitted (see section 6.5.2).
25. Concomitant or past history of psychiatric or neurologic disorder other than those considered to be related to AD (e.g., head injury with loss of consciousness, symptomatic stroke, Parkinson's disease, severe carotid occlusive disease, transient ischemic attacks, hemorrhagic and/or non-hemorrhagic stroke).
26. DSM-5 criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
27. Significant risk of suicide defined, using the C-SSRS, as the participant answering "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior within the past 6 months.
28. Clinically significant abnormal vital signs including sustained sitting blood pressure >160/90 mm Hg.
29. Participants with diabetes mellitus with hemoglobin A1c (HbA1c) levels of >7.5%.
30. In the opinion of the site PI, clinically significant deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, including, but not limited to:

    1. hematocrit less than 35% for those with male biological sex and less than 32% for those with female biological sex.
    2. absolute neutrophil cell count <1500/uL (with the exception of a chronic benign neutropenia).
    3. absolute lymphocyte count <900/uL.
    4. platelet cell count of <100,000/uL.
    5. INR >1.4 or other coagulopathy, confirmed by repeat (not applicable for participants on anticoagulation).
31. Participants with a known history of human immunodeficiency virus infection (HIV-1 and 2).
32. Participants with known history of acute/chronic hepatitis B or C.
33. Any other clinically significant, advanced, or unstable disease that may interfere with outcome evaluations, such as:

    1. Chronic liver disease.
    2. Respiratory insufficiency.
    3. Renal insufficiency defined as estimated glomerular filtration rate (eGFR) <50 mL/min based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
    4. Bradycardia (<50/min) or tachycardia (>100/min). Bradycardia >40/min and <50/min may be permitted with review and approval by the Medical Monitor.
34. Clinically significant arrhythmias or other clinically significant abnormalities on ECG at screening (minor abnormalities documented as clinically insignificant by the site PI are allowed).
35. Any condition, which in the opinion of the site PI, Coordinating Center, or Project Lead/Protocol PI, makes the participant unsuitable for inclusion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of brain tau deposition as measured by tau positron emission tomography (PET) | 0, 6, 18 and 30 months
  To determine whether at least one tau therapy, either alone or in combination with an anti-amyloid monoclonal antibody (mAb), will produce a greater reduction in brain tau deposition as measured by 18F-MK-6240 PET compared to anti-amyloid mAb alone.

SECONDARY OUTCOMES:
Disease progression as measured by plasma biomarkers | 30 months
  To assess whether at least one tau therapy, either alone or in combination with an anti-amyloid monoclonal antibody (mAb) slows disease progression as measured by plasma biomarkers. Plasma biomarkers are measured by the ratio of amyloid-beta 42 to amyloid-beta 40 (Aβ42/40), phosphorylated tau at threonine 217 (ptau217), neurofilament light chain (NfL), or glial fibrillary acid protein (GFAP).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco (UCSF), Memory and Aging Center; Keith Johnson, MD, Principal Investigator — Massachusetts General Hospital (MGH), Harvard Medical School

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: ACTC Alzheimer's Tau Platform — https://www.actcinfo.org/trial/alzheimers-tau-platform-atp-clinical-trial/